CLINICAL TRIAL: NCT05931354
Title: Longitudinal Study of Human Papillomavirus (HPV) Genotyping and Pap Smear in Patients With Antecedent Cervical Intraepithelial Neoplasia (CIN) and Association With Vaginal Intraepithelial Neoplasia (VAIN)
Brief Title: Longitudinal HPV Pap in CIN and VAIN
Acronym: LHPCV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201700471B0
Record Dates: First submitted 2023-06-27; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Cervical Intraepithelial Neoplasia; Hysterectomy; Human Papillomavirus; Vaginal Intraepithelial Neoplasia
Keywords: Cervical Intraepithelial Neoplasia; hysterectomy; human papillomavirus; vaginal intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Papanicolaou Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIN_Group: Those with a previous history of cervical cancer or CIN before incident VaIN and those with VaIN detected concomitantly with cervical cancer or CIN for whom both vaginal biopsy and cervical specimens were available in our hospital were eligible.
  Interventions: Other: HPV test and Pap Smear

INTERVENTIONS:
Other: HPV test and Pap Smear — HPV test and Pap Smear

SUMMARY:
This study will construct a longitudinal risk model of VaIN according to the HPVs distribution of cervix and vaginal for those had CIN2+. The study will include three arms to complete the follow-up data for the previous cohort constructed, and prospectively recruit new subjects with the appropriate inclusion/excluding criteria in order to increase sample size of this study.

DETAILED DESCRIPTION:
The long-term outcomes of patients with antecedent cervical intraepithelial neoplasia (CIN) were lacking. A systematic review published in 2008 identified no studies that met the review eligibility criteria for the prevalence of HPV types among vaginal precursors and cancers. Two sporadic studies containing 16 and 81 cases were reported in that review. Given that vaginal intraepithelial neoplasia (VAIN) post-hysterectomy for CIN is an uncommon disease which has a prevalence of being 1 to 6 %; it has the potential to progress to malignancy. Although the etiology of VAIN has not been as thoroughly investigated as that of CIN, evidence implicates that the human papillomavirus (HPV) as the probable carcinogenic agent for the onset and evolution of some VAIN and vaginal cancers.

This study will construct a longitudinal risk model of VaIN according to the HPVs distribution of cervix and vaginal for those had CIN2+.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 20 years
2. Those with a previous history of CIN+

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with a previous history of cervical cancer or CIN before incident VaIN and those with VaIN detected concomitantly with cervical cancer or CIN for whom both vaginal biopsy and cervical specimens
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
progression rate of CIN+ or VaIN+ | 5 years
  time to developing CIN+ or VaIN+ from first CIN+ diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Medical Foundation, Taoyuan, Taiwan